CLINICAL TRIAL: NCT02223832
Title: Single-center, Open-label, Parallel-group Study to Evaluate the Pharmacokinetics, Tolerability, and Safety of a Single Dose of 40 mg ACT-128800 in Japanese and Caucasian Healthy Male and Female Subjects
Brief Title: Study to Evaluate the Pharmacokinetics, Tolerability, and Safety of ACT-128800 in Japanese and Caucasian Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AC-058-107
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: ACT-128800; Safety; Tolerability; Pharmacokinetics
MeSH Terms: interventions — ponesimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACT-128800 (Experimental): A single oral dose of 40 mg ACT-128800 will be administered as
  1 capsule given in the fasted state in the morning
  Interventions: Drug: ACT-128800

INTERVENTIONS:
Drug: ACT-128800

SUMMARY:
This is a study to evaluate the relative pharmacokinetic properties and the tolerability and safety of ACT-128800 in Japanese and Caucasian healthy male and female subjects after single-dose administration.

DETAILED DESCRIPTION:
10 Japanese and 10 Caucasian healthy male and female subjects in a one to one male to female ratio will be included in the study. Japanese and Caucasian subjects will be matched for body weight.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Japanese or Caucasian. (Japanese subjects: both parents of the subject are Japanese [born in Japan]. Caucasian subjects: both parents of the subject are Caucasian).
* Body mass index between 18 and 28 kg/m^2, inclusive.
* Women not of childbearing potential:
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to drug intake on Day 1; use a reliable method of contraception and continue this contraception for the duration of the study and for at least 2 months after study drug intake. In addition, her partner must use a condom.
* Systolic blood pressure 100-145 mmHg, diastolic blood pressure 50-90 mmHg, and heart rate (HR) 50-95 beats per minute (inclusive).
* 12-lead electrocardiogram without clinically relevant abnormalities at screening.
* Hematology and clinical chemistry results not deviating from the normal range to a clinically relevant extent at screening.
* Negative results from urine drug screen at screening.
* Ability to communicate well with the Investigator (if necessary with the help of an interpreter) and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Electrocardiograph PQ/PR interval (time interval from the beginning of the P wave to the beginning of the QRS complex) > 200 milliseconds at screening.
* Nursing woman.
* History of asthma or chronic obstructive pulmonary disease.
* Known hypersensitivity to any excipients of the drug formulation.
* Treatment with another investigational drug within 3 months prior to screening.
* Excessive caffeine consumption, defined as > 800 mg per day at screening.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition that might interfere with the absorption, distribution, metabolism or excretion of the study drug.
* Any cardiac condition or illness, including ECG abnormalities, with a potential to increase the cardiac risk of the subject.
* Smoking within the last month prior to screening.
* Any immunosuppressive treatment within 6 weeks before study drug administration.
* Previous treatment with any prescribed or over-the-counter medications within 2 weeks prior to screening.
* Loss of 250 mL or more of blood within 3 months prior to screening.
* Lymphopenia (< 1,000 lymphocytes/μL).
* Viral, fungal, bacterial or protozoal infection within 4 weeks before study drug administration.
* Positive results from the hepatitis serology, except for vaccinated subjects, at screening.
* Positive results from human immunodeficiency vrus serology at screening.
* Legal incapacity or limited legal capacity at screening.
* History of alcoholism or drug abuse.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure from baseline up to end of study | Up to 10 days
  Blood pressure shall be measured using an automatic oscillometric device, always on the leading (writing) arm. Measurements shall be taken in the supine position after having rested for at least a 5 min period.
Change in diastolic blood pressure from baseline up to end of study | Up to 10 days
  Blood pressure shall be measured using an automatic oscillometric device, always on the leading (writing) arm. Measurements shall be taken in the supine position after having rested for at least a 5 min period.
Change in pulse rate from baseline up to end of study | Up to 10 days
  Pulse rate shall be measured using an automatic oscillometric device, always on the leading (writing) arm. Measurements shall be taken in the supine position after having rested for at least a 5 min period.
Change in body temperature from baseline up to end of study | Up to 10 days
  Body temperature shall be measured in a supine position using the same thermometer throughout the study.
Change in forced expiratory volume in 1 second (FEV1) from baseline up to end of study | Up to 10 days
  FEV1 assessments shall be performed in a standardized manner as per the American Thoracic Society standards. Three good test breaths will be measured; the highest FEV1 value from these three breath tests will be recorded.
Change in forced vital capacity (FVC) from baseline up to end of study | Up to 10 days
  FVC assessments shall be performed in a standardized manner as per the American Thoracic Society standards. Three good test breaths will be measured; the highest FVC value from these three breath tests will be recorded.
Number of treatment-emergent abnormalities on physical examination up to end of study | Up to 10 days
  Physical examination (i.e., inspection, percussion, palpation, and auscultation) shall be performed during the course of the study.
Change in heart rate from baseline up to end of study | Up to 10 days
  Heart rate shall be measured using standard 12-lead electrocardiogram recorded at rest with the subject in the supine position for a 5-minute period.
Change in QT interval (time interval from beginning of the Q wave until end of the T wave) calculated according to Bazett's correction (QTcB) from baseline up to end of study | Up to 10 days
  QTcB shall be determined using standard 12-lead electrocardiogram recorded at rest with the subject in the supine position for a 5-minute period. The QTcB interval is the QT interval corrected for heart rate with Bazett's formula (QTcB = QT/RR^0.5 where RR is 60/heart rate).
Change in QT interval (time interval from beginning of the Q wave until end of the T wave) calculated according to Fridericia's correction (QTcF) from baseline up to end of study | Up to 10 days
  QTcF shall be determined using standard 12-lead electrocardiogram recorded at rest with the subject in the supine position for a 5-minute period. The QTcF interval is the QT interval corrected for heart rate with Fridericia's formula (QTcF = QT/RR^0.33 where RR is 60/heart rate).
Number of treatment-emergent electrocardiogram abnormalities up to end of study | Up to 10 days
  Electrocardiogram abnormalities shall be determined using standard 12-lead electrocardiogram recorded at rest with the subject in the supine position for a 5-minute period.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of ACT-128800 | 144 hours
  Blood samples for pharmacokinetic analysis shall be taken immediately prior to dosing with ACT-128800 and at 0.5, 1, 1.5, 2.5, 4, 6, 10, 16, 24, 36, 48, 72, 96, 120 and 144 hours after dosing. Cmax will be calculated on the basis of the blood sampling time points.
Time to maximum plasma concentration (tmax) of ACT-128800 | 144 hours
  Blood samples for pharmacokinetic analysis shall be taken immediately prior to dosing with ACT-128800 and at 0.5, 1, 1.5, 2.5, 4, 6, 10, 16, 24, 36, 48, 72, 96, 120 and 144 hours after dosing. tmax will be calculated on the basis of the blood sampling time points.
Area under the plasma concentration-time curve (AUC(0-t)) of ACT-128800 | 144 hours
  Blood samples for pharmacokinetic analysis shall be taken immediately prior to dosing with ACT-128800 and at 0.5, 1, 1.5, 2.5, 4, 6, 10, 16, 24, 36, 48, 72, 96, 120 and 144 hours after dosing. AUC(0-t) shall be calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification
Area under the plasma concentration-time curve (AUC(0-infinity)) of ACT-128800 | 144 hours
  Blood samples for pharmacokinetic analysis shall be taken immediately prior to dosing with ACT-128800 and at 0.5, 1, 1.5, 2.5, 4, 6, 10, 16, 24, 36, 48, 72, 96, 120 and 144 hours after dosing. AUC(0-infinity) will be calculated by combining AUC(0-t) and AUC(extra). AUC(extra) represents an extrapolated value obtained by Ct/λZ, where Ct is the last plasma concentration measured above the limit of quantification and λZ represents the terminal elimination rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal elimination phase.
Plasma half life (t1/2) of ACT-128800 | 144 hours
  Blood samples for pharmacokinetic analysis shall be taken immediately prior to dosing with ACT-128800 and at 0.5, 1, 1.5, 2.5, 4, 6, 10, 16, 24, 36, 48, 72, 96, 120 and 144 hours after dosing. t1/2 will be calculated on the basis of the blood sampling time points.
Change in lymphocyte count from baseline up to end of study | Up to 10 days
  At various time points up to the end of study about 3 mL of blood will be collected by venepuncture in the supine position, for the measurement of lymphocyte count.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Brossard, PhD, Study Director — Actelion Pharmaceuticals Limited
Locations (1):
- Hawaii Clinical Research Center, Honolulu, Hawaii, United States